CLINICAL TRIAL: NCT06295250
Title: ASHA Bangladesh--An Integrated Intervention to Address Depression in Low Income Rural Women
Brief Title: ASHA Bangladesh--An Integrated Intervention to Address Poverty and Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Georgetown University (Other); National Institute of Mental Health (NIMH) (NIH); Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Alison Karasz, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00001114; 7R01MH127577 (NIH)
Record Dates: First submitted 2024-02-27; First posted 2024-03-06 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Depression; Economic Vulnerability
Keywords: Depression treatment; Cash Transfer; Problem Management Plus; Poverty Alleviation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Blinding is difficult with behavioral studies. In this trial, efforts will be made to keep participants and interventionists from learning details of the trial design and alternate interventions. Outcome assessors will be blinded to randomization assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Depression Treatment (DT) (Active Comparator): Participants in the control group will receive a 10 session 6 month manualized group based psychotherapy treatment..
  Interventions: Behavioral: Manualized Group Based Psychotherapy
- Integrated Intervention (Experimental): The experimental arm includes 2 elements:
  1. The psychotherapy intervention described above.
  2. A poverty alleviation intervention
  Interventions: Behavioral: Manualized Group Based Psychotherapy; Other: Poverty Alleviation

INTERVENTIONS:
Behavioral: Manualized Group Based Psychotherapy — Manualized Group Based Psychotherapy. Adapted from the World Health Organization (WHO) Problem Management Plus (PM+) intervention, this intervention includes behavioral activation, enhancing social support, and problem management.
Other: Poverty Alleviation — Modeled on the well-known Graduation Program, a poverty alleviation strategy widely used in low income countries, this intervention includes an asset transfer (agricultural animals), financial literacy education, a 6 month stipend, savings accounts, veterinary support, feed, and agricultural training
  Arms: Integrated Intervention

SUMMARY:
The goal of this randomized controlled trial is to compare the impact of an integrated intervention combining poverty alleviation and depression treatment to depression treatment alone, in low income rural Bangladeshi women with depression. The main question[s] it aims to answer are whether adding poverty alleviation to depression treatment in an integrated intervention: 1) improves depression outcomes at 6 months post baseline as measured by changes in the PHQ-9 from baseline; 2) reduces the chance of relapse (PHQ-9 >=10) at 24 months among patients who remitted (PHQ-9>=5) at six months; and 2) whether adding poverty alleviation to depression treatment improves implementation outcomes including treatment uptake and retention. Participants in both arms will participate in research interviews at 6,12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. married women;
2. age 18-75;
3. fluent in Bengali);
4. Meets criteria on an Economic Vulnerability Index
5. >=10 on the Patient Health Questionnaire (PHQ-9 Depression Scale at baseline

Exclusion Criteria:

1. Inability to provide informed consent;
2. Plans to travel for > 1 month during 24 M period.
3. Inability to participate in the study for any other reason

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change in Depressive symptoms at 6 Months | 6 Months
  Change in Symptoms from Baseline to 6 months post baseline, as measured by the Patient Health Questionnaire, a 9 item questionnaire designed to assess depressive symptoms. The minimum score is 0; the maximum score is 27.
24 Month Relapse | 24 months
  Relapse is defined as a score of Patient Health Questionnaire>= 10 among participants who achieved remission at Time 2--6 months. To assess relapse, at each data collection point (6, 12, and 24 month) the investigators will ask participants about the experience of depressive symptoms at any time since the previous data collection point. Data collection will focus on 24 month relapse, or the presence of relapse at any time since Time 2.

SECONDARY OUTCOMES:
Economic vulnerability index | Baseline, 12, and 24 Months
  A composite index of economic vulnerability that includes income, assets, debt, food insecurity, financial worry. This measure does not have a fixed score but is composed using a pragmatic approach based on data collected in the field.
Anxiety | Baseline, 6 Months, 12 Months, and 24 Months
  Anxiety symptoms as measured on the General Anxiety Disorder scale--a seven item questionnaire with scores from 0-231. HIgher scores indicate more anxiety.
Function | Baseline, 6 Months, 12 Months, and 24 Months
  Function and disability as measured by the World Health Organization Disability Assessment Schedule, a 12 item questionnaire that is scored from 12-60 with higher scores indicating greater disability.
Change in Quality of Life | Baseline, 6 Months, 12 Months, and 24 Months
  Quality of life measure that includes five dimensions: mobility, self care, usual activities, pain/discomfort and anxiety/depression, scored from 0-100 with higher scores indicating better quality of life.
Tension Scale | Baseline, 6 Months, 12 Months, 18 months and 24 Months
  A questionnaire that measures both psychological symptoms as well as somatic cultural symptoms: a 39 item instrument measured from 0-3 with a minimum score of 0 and a maximum score of 117. with higher scores indicating higher levels of distress.

OTHER OUTCOMES:
Implementation Outcomes--Adoption | Baseline + 30 days
  The number of participants attending >-1 treatment session/# participants randomized. Based on recruitment and study records.
Implementation Outcomes--Feasibility | Six months
  Percent of participants attending >= 75 percent of intervention sessions--based on study records
Implementation outcomes--fidelity | Intervention months 1, 3 and 6
  Supervisor observations of sessions will be assessed for fidelity using a LIKERT scale that includes preparedness (0-3), Facilitation (0-11), Engagement (0-6) time management (0-1) and Documentation (0-1).

CONTACTS AND LOCATIONS:
Overall Officials: Alison Karasz, PhD, Principal Investigator — UMass Chan Medical School
Locations (1):
- International Centre for Diarrhoeal Disease Research, Dhaka, Dhaka Division, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
We will create a deidentified dataset and it is our intention that these data be readily accessible and used. We will collaborate with and make our data available to other researchers for additional/secondary analyses. Formal data sharing agreements will be developed to guide and encourage further data mining of the proposed datasets for various purposes. All such data requests will be approved though by the investigative team, including the International Center for Diarrhoeal Disease Research (ICDDRB), to help ensure ethical use of the data.
Supporting Information: Analytic Code
Time Frame: Data will be available indefinitely following the completion of analyses
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Background] Greenberg PE, Kessler RC, Birnbaum HG, Leong SA, Lowe SW, Berglund PA, Corey-Lisle PK. The economic burden of depression in the United States: how did it change between 1990 and 2000? J Clin Psychiatry. 2003 Dec;64(12):1465-75. doi: 10.4088/jcp.v64n1211. PMID 14728109
- [Background] Kessler RC, Akiskal HS, Ames M, Birnbaum H, Greenberg P, Hirschfeld RM, Jin R, Merikangas KR, Simon GE, Wang PS. Prevalence and effects of mood disorders on work performance in a nationally representative sample of U.S. workers. Am J Psychiatry. 2006 Sep;163(9):1561-8. doi: 10.1176/ajp.2006.163.9.1561. PMID 16946181
- [Background] Heflin CM, Iceland J. Poverty, Material Hardship and Depression. Soc Sci Q. 2009 Dec 1;90(5):1051-1071. doi: 10.1111/j.1540-6237.2009.00645.x. PMID 25530634
- [Background] Haushofer J, Fehr E. On the psychology of poverty. Science. 2014 May 23;344(6186):862-7. doi: 10.1126/science.1232491. PMID 24855262
- [Background] Patel V, Araya R, de Lima M, Ludermir A, Todd C. Women, poverty and common mental disorders in four restructuring societies. Soc Sci Med. 1999 Dec;49(11):1461-71. doi: 10.1016/s0277-9536(99)00208-7. PMID 10515629
- [Background] Lerman S. The syndemogenesis of depression Concepts and examples. depression. 2018.
- [Background] Lund C, De Silva M, Plagerson S, Cooper S, Chisholm D, Das J, Knapp M, Patel V. Poverty and mental disorders: breaking the cycle in low-income and middle-income countries. Lancet. 2011 Oct 22;378(9801):1502-14. doi: 10.1016/S0140-6736(11)60754-X. Epub 2011 Oct 16. PMID 22008425
- [Background] Lund C, Breen A, Flisher AJ, Kakuma R, Corrigall J, Joska JA, Swartz L, Patel V. Poverty and common mental disorders in low and middle income countries: A systematic review. Soc Sci Med. 2010 Aug;71(3):517-528. doi: 10.1016/j.socscimed.2010.04.027. Epub 2010 May 12. PMID 20621748
- [Background] Program UND. Human development report 2019: Beyond income, beyond averages, beyond today: Inequalities in human development in the 21st century. 2019.
- [Background] Buckshee K. Impact of roles of women on health in India. Int J Gynaecol Obstet. 1997 Jul;58(1):35-42. doi: 10.1016/s0020-7292(97)02887-7. PMID 9253664
- [Background] Jambunathan J. Sociocultural factors in depression in Asian Indian women. Health Care Women Int. 1992 Jul-Sep;13(3):261-70. doi: 10.1080/07399339209516001. PMID 1399866
- [Background] Rani M, Bonu S. Rural Indian women's care-seeking behavior and choice of provider for gynecological symptoms. Stud Fam Plann. 2003 Sep;34(3):173-85. doi: 10.1111/j.1728-4465.2003.00173.x. PMID 14558320
- [Background] Rodrigues M, Patel V, Jaswal S, de Souza N. Listening to mothers: qualitative studies on motherhood and depression from Goa, India. Soc Sci Med. 2003 Nov;57(10):1797-806. doi: 10.1016/s0277-9536(03)00062-5. PMID 14499506
- [Background] Ullrich HE. A study of change and depression among Havik Brahmin women in a south Indian village. Cult Med Psychiatry. 1987 Sep;11(3):261-87. doi: 10.1007/BF00048516. PMID 3677776
- [Background] Karasz A. Marriage, Depression and Illness: Sociosomatic Models in a South Asian Immigrant Community. Psychology and Developing Societies. 2005;17(2):161-180.
- [Background] Sparling TM, Waid JL, Wendt AS, Gabrysch S. Depression among women of reproductive age in rural Bangladesh is linked to food security, diets and nutrition. Public Health Nutr. 2020 Mar;23(4):660-673. doi: 10.1017/S1368980019003495. Epub 2020 Jan 9. PMID 31915095
- [Background] Rahman A, Patel V, Maselko J, Kirkwood B. The neglected 'm' in MCH programmes--why mental health of mothers is important for child nutrition. Trop Med Int Health. 2008 Apr;13(4):579-83. doi: 10.1111/j.1365-3156.2008.02036.x. Epub 2008 Mar 3. PMID 18318697
- [Background] Harpham T, Huttly S, De Silva MJ, Abramsky T. Maternal mental health and child nutritional status in four developing countries. J Epidemiol Community Health. 2005 Dec;59(12):1060-4. doi: 10.1136/jech.2005.039180. PMID 16286495
- [Background] Nguyen PH, Saha KK, Ali D, Menon P, Manohar S, Mai LT, Rawat R, Ruel MT. Maternal mental health is associated with child undernutrition and illness in Bangladesh, Vietnam and Ethiopia. Public Health Nutr. 2014 Jun;17(6):1318-27. doi: 10.1017/S1368980013001043. Epub 2013 May 3. PMID 23642497
- [Background] Sharmin KN, Sarwar N, Mumu SJ, Taleb DA, Flora MS. Postnatal depression and infant growth in an urban area of Bangladesh. Midwifery. 2019 Jul;74:57-67. doi: 10.1016/j.midw.2019.03.014. Epub 2019 Mar 22. PMID 30927633
- [Background] Nyatsanza M, Schneider M, Davies T, Lund C. Filling the treatment gap: developing a task sharing counselling intervention for perinatal depression in Khayelitsha, South Africa. BMC Psychiatry. 2016 May 26;16:164. doi: 10.1186/s12888-016-0873-y. PMID 27228979
- [Background] Patel V, Rodrigues M, DeSouza N. Gender, poverty, and postnatal depression: a study of mothers in Goa, India. Am J Psychiatry. 2002 Jan;159(1):43-7. doi: 10.1176/appi.ajp.159.1.43. PMID 11772688
- [Background] Patel V, Saraceno B, Kleinman A. Beyond evidence: the moral case for international mental health. Am J Psychiatry. 2006 Aug;163(8):1312-5. doi: 10.1176/ajp.2006.163.8.1312. No abstract available. PMID 16877638
- [Background] Patel V, Simon G, Chowdhary N, Kaaya S, Araya R. Packages of care for depression in low- and middle-income countries. PLoS Med. 2009 Oct;6(10):e1000159. doi: 10.1371/journal.pmed.1000159. Epub 2009 Oct 6. PMID 19806179
- [Background] Patel V, Prince M. Global mental health: a new global health field comes of age. JAMA. 2010 May 19;303(19):1976-7. doi: 10.1001/jama.2010.616. No abstract available. PMID 20483977
- [Background] Patel V, Chowdhary N, Rahman A, Verdeli H. Improving access to psychological treatments: lessons from developing countries. Behav Res Ther. 2011 Sep;49(9):523-8. doi: 10.1016/j.brat.2011.06.012. Epub 2011 Jul 7. PMID 21788012
- [Background] Patel V, Collins PY, Copeland J, Kakuma R, Katontoka S, Lamichhane J, Naik S, Skeen S. The movement for global mental health. Br J Psychiatry. 2011 Feb;198(2):88-90. doi: 10.1192/bjp.bp.109.074518. PMID 21282777
- [Background] Rajaraman D, Travasso S, Chatterjee A, Bhat B, Andrew G, Parab S, Patel V. The acceptability, feasibility and impact of a lay health counsellor delivered health promoting schools programme in India: a case study evaluation. BMC Health Serv Res. 2012 May 25;12:127. doi: 10.1186/1472-6963-12-127. PMID 22630607
- [Background] Shinde S, Andrew G, Bangash O, Cohen A, Kirkwood B, Patel V. The impact of a lay counselor led collaborative care intervention for common mental disorders in public and private primary care: a qualitative evaluation nested in the MANAS trial in Goa, India. Soc Sci Med. 2013 Jul;88:48-55. doi: 10.1016/j.socscimed.2013.04.002. Epub 2013 Apr 9. PMID 23702209
- [Background] Cuijpers P, Karyotaki E, Reijnders M, Purgato M, Barbui C. Psychotherapies for depression in low- and middle-income countries: a meta-analysis. World Psychiatry. 2018 Feb;17(1):90-101. doi: 10.1002/wps.20493. PMID 29352530
- [Background] Rahman A, Fisher J, Bower P, Luchters S, Tran T, Yasamy MT, Saxena S, Waheed W. Interventions for common perinatal mental disorders in women in low- and middle-income countries: a systematic review and meta-analysis. Bull World Health Organ. 2013 Aug 1;91(8):593-601I. doi: 10.2471/BLT.12.109819. Epub 2013 Apr 18. PMID 23940407
- [Background] Shidhaye R, Baron E, Murhar V, Rathod S, Khan A, Singh A, Shrivastava S, Muke S, Shrivastava R, Lund C, Patel V. Community, facility and individual level impact of integrating mental health screening and treatment into the primary healthcare system in Sehore district, Madhya Pradesh, India. BMJ Glob Health. 2019 May 19;4(3):e001344. doi: 10.1136/bmjgh-2018-001344. eCollection 2019. PMID 31179034
- [Background] Sikander S, Ahmad I, Atif N, Zaidi A, Vanobberghen F, Weiss HA, Nisar A, Tabana H, Ain QU, Bibi A, Bilal S, Bibi T, Liaqat R, Sharif M, Zulfiqar S, Fuhr DC, Price LN, Patel V, Rahman A. Delivering the Thinking Healthy Programme for perinatal depression through volunteer peers: a cluster randomised controlled trial in Pakistan. Lancet Psychiatry. 2019 Feb;6(2):128-139. doi: 10.1016/S2215-0366(18)30467-X. PMID 30686386
- [Background] Fuhr DC, Weobong B, Lazarus A, Vanobberghen F, Weiss HA, Singla DR, Tabana H, Afonso E, De Sa A, D'Souza E, Joshi A, Korgaonkar P, Krishna R, Price LN, Rahman A, Patel V. Delivering the Thinking Healthy Programme for perinatal depression through peers: an individually randomised controlled trial in India. Lancet Psychiatry. 2019 Feb;6(2):115-127. doi: 10.1016/S2215-0366(18)30466-8. PMID 30686385
- [Background] Patel V, Weiss HA, Chowdhary N, Naik S, Pednekar S, Chatterjee S, De Silva MJ, Bhat B, Araya R, King M, Simon G, Verdeli H, Kirkwood BR. Effectiveness of an intervention led by lay health counsellors for depressive and anxiety disorders in primary care in Goa, India (MANAS): a cluster randomised controlled trial. Lancet. 2010 Dec 18;376(9758):2086-95. doi: 10.1016/S0140-6736(10)61508-5. Epub 2010 Dec 13. PMID 21159375
- [Background] Lund C, Schneider M, Garman EC, Davies T, Munodawafa M, Honikman S, Bhana A, Bass J, Bolton P, Dewey M, Joska J, Kagee A, Myer L, Petersen I, Prince M, Stein DJ, Tabana H, Thornicroft G, Tomlinson M, Hanlon C, Alem A, Susser E. Task-sharing of psychological treatment for antenatal depression in Khayelitsha, South Africa: Effects on antenatal and postnatal outcomes in an individual randomised controlled trial. Behav Res Ther. 2020 Jul;130:103466. doi: 10.1016/j.brat.2019.103466. Epub 2019 Oct 31. PMID 31733813
- [Background] Westen D, Novotny CM, Thompson-Brenner H. The empirical status of empirically supported psychotherapies: assumptions, findings, and reporting in controlled clinical trials. Psychol Bull. 2004 Jul;130(4):631-63. doi: 10.1037/0033-2909.130.4.631. PMID 15250817
- [Background] Thase ME, Simons AD, McGeary J, Cahalane JF, Hughes C, Harden T, Friedman E. Relapse after cognitive behavior therapy of depression: potential implications for longer courses of treatment. Am J Psychiatry. 1992 Aug;149(8):1046-52. doi: 10.1176/ajp.149.8.1046. PMID 1636804
- [Background] Leichsenring F, Rabung S. Effectiveness of long-term psychodynamic psychotherapy: a meta-analysis. JAMA. 2008 Oct 1;300(13):1551-65. doi: 10.1001/jama.300.13.1551. PMID 18827212
- [Background] Leichsenring F, Rabung S. Long-term psychodynamic psychotherapy in complex mental disorders: update of a meta-analysis. Br J Psychiatry. 2011 Jul;199(1):15-22. doi: 10.1192/bjp.bp.110.082776. PMID 21719877
- [Background] Warden D, Rush AJ, Wisniewski SR, Lesser IM, Thase ME, Balasubramani GK, Shores-Wilson K, Nierenberg AA, Trivedi MH. Income and attrition in the treatment of depression: a STAR*D report. Depress Anxiety. 2009;26(7):622-33. doi: 10.1002/da.20541. PMID 19582825
- [Background] Miranda J, Chung JY, Green BL, Krupnick J, Siddique J, Revicki DA, Belin T. Treating depression in predominantly low-income young minority women: a randomized controlled trial. JAMA. 2003 Jul 2;290(1):57-65. doi: 10.1001/jama.290.1.57. PMID 12837712
- [Background] Karasz A, Raghavan S, Patel V, Zaman M, Akhter L, Kabita M. ASHA: Using Participatory Methods to Develop an Asset-building Mental Health Intervention for Bangladeshi Immigrant Women. Prog Community Health Partnersh. 2015 Winter;9(4):501-12. doi: 10.1353/cpr.2015.0080. PMID 26639376
- [Background] Karasz A. Cultural differences in conceptual models of depression. Soc Sci Med. 2005 Apr;60(7):1625-35. doi: 10.1016/j.socscimed.2004.08.011. PMID 15652693
- [Background] Karasz A, Dempsey K. Health seeking for ambiguous symptoms in two cultural groups: a comparative study. Transcult Psychiatry. 2008 Sep;45(3):415-38. doi: 10.1177/1363461508094674. PMID 18799641
- [Background] Karasz A, Garcia N, Ferri L. Conceptual Models of Depression in Primary Care Patients: A Comparative Study. J Cross Cult Psychol. 2009 Nov 1;40(6):1041-1059. doi: 10.1177/0022022109348782. PMID 20182550
- [Background] Karasz A, Sacajiu G, Garcia N. Conceptual models of psychological distress among low-income patients in an inner-city primary care clinic. J Gen Intern Med. 2003 Jun;18(6):475-7. doi: 10.1046/j.1525-1497.2003.20636.x. PMID 12823655
- [Background] Karasz A, Watkins L. Conceptual models of treatment in depressed Hispanic patients. Ann Fam Med. 2006 Nov-Dec;4(6):527-33. doi: 10.1370/afm.579. PMID 17148631
- [Background] Aggarwal NK, Balaji M, Kumar S, Mohanraj R, Rahman A, Verdeli H, Araya R, Jordans MJ, Chowdhary N, Patel V. Using consumer perspectives to inform the cultural adaptation of psychological treatments for depression: a mixed methods study from South Asia. J Affect Disord. 2014 Jul;163(100):88-101. doi: 10.1016/j.jad.2014.03.036. Epub 2014 Apr 1. PMID 24836093
- [Background] Bhattacharya A, Camacho D, Kimberly LL, Lukens EP. Women's Experiences and Perceptions of Depression in India: A Metaethnography. Qual Health Res. 2019 Jan;29(1):80-95. doi: 10.1177/1049732318811702. PMID 30799765
- [Background] Roberts T, Shrivastava R, Koschorke M, Patel V, Shidhaye R, Rathod SD. "Is there a medicine for these tensions?" Barriers to treatment-seeking for depressive symptoms in rural India: A qualitative study. Soc Sci Med. 2020 Feb;246:112741. doi: 10.1016/j.socscimed.2019.112741. Epub 2019 Dec 19. PMID 31918347
- [Background] Karasz A. The development of valid subtypes for depression in primary care settings: a preliminary study using an explanatory model approach. J Nerv Ment Dis. 2008 Apr;196(4):289-96. doi: 10.1097/NMD.0b013e31816a496e. PMID 18414123
- [Background] Karasz A, Patel V, Kabita M, Shimu P. "Tension" in South Asian women: developing a measure of common mental disorder using participatory methods. Prog Community Health Partnersh. 2013 Winter;7(4):429-41. doi: 10.1353/cpr.2013.0046. PMID 24375184
- [Background] Grote NK, Zuckoff A, Swartz H, Bledsoe SE, Geibel S. Engaging women who are depressed and economically disadvantaged in mental health treatment. Soc Work. 2007 Oct;52(4):295-308. doi: 10.1093/sw/52.4.295. PMID 18232240
- [Background] Anderson CM, Robins CS, Greeno CG, Cahalane H, Copeland VC, Andrews RM. Why lower income mothers do not engage with the formal mental health care system: perceived barriers to care. Qual Health Res. 2006 Sep;16(7):926-43. doi: 10.1177/1049732306289224. PMID 16894224
- [Background] Schraufnagel TJ, Wagner AW, Miranda J, Roy-Byrne PP. Treating minority patients with depression and anxiety: what does the evidence tell us? Gen Hosp Psychiatry. 2006 Jan-Feb;28(1):27-36. doi: 10.1016/j.genhosppsych.2005.07.002. PMID 16377362
- [Background] Brown GW, Harris TO, Kendrick T, Chatwin J, Craig TK, Kelly V, Mander H, Ring A, Wallace V, Uher R; Thread Study Group. Antidepressants, social adversity and outcome of depression in general practice. J Affect Disord. 2010 Mar;121(3):239-46. doi: 10.1016/j.jad.2009.06.004. Epub 2009 Jul 9. PMID 19589602
- [Background] Jakubovski E, Bloch MH. Prognostic subgroups for citalopram response in the STAR*D trial. J Clin Psychiatry. 2014 Jul;75(7):738-47. doi: 10.4088/JCP.13m08727. PMID 24912106
- [Background] Zayas LH, McKee MD, Jankowski KR. Adapting psychosocial intervention research to urban primary care environments: a case example. Ann Fam Med. 2004 Sep-Oct;2(5):504-8. doi: 10.1370/afm.108. PMID 15506589
- [Background] Falconnier L. Socioeconomic status in the treatment of depression. Am J Orthopsychiatry. 2009 Apr;79(2):148-58. doi: 10.1037/a0015469. PMID 19485632
- [Background] Cohen A, Gilman SE, Houck PR, Szanto K, Reynolds CF 3rd. Socioeconomic status and anxiety as predictors of antidepressant treatment response and suicidal ideation in older adults. Soc Psychiatry Psychiatr Epidemiol. 2009 Apr;44(4):272-7. doi: 10.1007/s00127-008-0436-8. Epub 2008 Sep 25. PMID 18818858
- [Background] Cohen A, Houck PR, Szanto K, Dew MA, Gilman SE, Reynolds CF 3rd. Social inequalities in response to antidepressant treatment in older adults. Arch Gen Psychiatry. 2006 Jan;63(1):50-6. doi: 10.1001/archpsyc.63.1.50. PMID 16389196
- [Background] Jain FA, Hunter AM, Brooks JO 3rd, Leuchter AF. Predictive socioeconomic and clinical profiles of antidepressant response and remission. Depress Anxiety. 2013 Jul;30(7):624-30. doi: 10.1002/da.22045. Epub 2013 Jan 3. PMID 23288666
- [Background] Conradi HJ, Bos EH, Kamphuis JH, de Jonge P. The ten-year course of depression in primary care and long-term effects of psychoeducation, psychiatric consultation and cognitive behavioral therapy. J Affect Disord. 2017 Aug 1;217:174-182. doi: 10.1016/j.jad.2017.03.064. Epub 2017 Mar 30. PMID 28411506
- [Background] van Weel-Baumgarten EM, Schers HJ, van den Bosch WJ, van den Hoogen HJ, Zitman FG. Long-term follow-up of depression among patients in the community and in family practice settings. A systematic review. J Fam Pract. 2000 Dec;49(12):1113-20. PMID 11132061
- [Background] Brugha TS, Bebbington PE, MacCarthy B, Sturt E, Wykes T. Antidepressants may not assist recovery in practice: a naturalistic prospective survey. Acta Psychiatr Scand. 1992 Jul;86(1):5-11. doi: 10.1111/j.1600-0447.1992.tb03218.x. PMID 1414401
- [Background] Johansson O, Lundh LG, Bjarehed J. 12-Month Outcome and Predictors of Recurrence in Psychiatric Treatment of Depression: A Retrospective Study. Psychiatr Q. 2015 Sep;86(3):407-17. doi: 10.1007/s11126-015-9341-y. PMID 25597030
- [Background] Steinert C, Hofmann M, Kruse J, Leichsenring F. Relapse rates after psychotherapy for depression - stable long-term effects? A meta-analysis. J Affect Disord. 2014 Oct;168:107-18. doi: 10.1016/j.jad.2014.06.043. Epub 2014 Jul 2. PMID 25043322
- [Background] Vittengl JR, Jarrett RB. Cognitive Therapy to Prevent Depressive Relapse in Adults. Curr Opin Psychol. 2015 Aug 1;4:26-31. doi: 10.1016/j.copsyc.2015.01.016. PMID 25729758
- [Background] Haushofer J, Mudida R, Shapiro J. The Comparative Impact of Cash Transfers and Psychotherapy on Psychological and Economic Well-being. 2019.
- [Background] Burgess R, Campbell C. Contextualising women's mental distress and coping strategies in the time of AIDS: a rural South African case study. Transcult Psychiatry. 2014 Dec;51(6):875-903. doi: 10.1177/1363461514526925. Epub 2014 Mar 26. PMID 24670517
- [Background] Summerfield D. How scientifically valid is the knowledge base of global mental health? BMJ. 2008 May 3;336(7651):992-4. doi: 10.1136/bmj.39513.441030.AD. PMID 18456630
- [Background] Grote NK, Swartz HA, Zuckoff A. Enhancing Interpersonal Psychotherapy for Mothers and Expectant Mothers on Low Incomes: Adaptations and Additions. J Contemp Psychother. 2008 Mar;38(1):23-33. doi: 10.1007/s10879-007-9065-x. PMID 21822328
- [Background] Patel V, Burns JK, Dhingra M, Tarver L, Kohrt BA, Lund C. Income inequality and depression: a systematic review and meta-analysis of the association and a scoping review of mechanisms. World Psychiatry. 2018 Feb;17(1):76-89. doi: 10.1002/wps.20492. PMID 29352539
- [Background] Weber H. The 'new economy' and social risk: banking on the poor? Review of International Political Economy. 2004;11(2):356-386.
- [Background] Murshid NS, Akincigil A, Zippay A. Microfinance Participation and Domestic Violence in Bangladesh: Results From a Nationally Representative Survey. J Interpers Violence. 2016 May;31(9):1579-96. doi: 10.1177/0886260515569065. Epub 2015 Feb 4. PMID 25657103
- [Background] Hunt J, Kasynathan N. Pathways to empowerment? Reflections on microfinance and transformation in gender relations in South Asia. Gender & Development. 2001;9(1):42-52.
- [Background] Baird SJ, Garfein RS, McIntosh CT, Ozler B. Effect of a cash transfer programme for schooling on prevalence of HIV and herpes simplex type 2 in Malawi: a cluster randomised trial. Lancet. 2012 Apr 7;379(9823):1320-9. doi: 10.1016/S0140-6736(11)61709-1. Epub 2012 Feb 15. PMID 22341825
- [Background] Banerjee A, Duflo E, Goldberg N, Karlan D, Osei R, Pariente W, Shapiro J, Thuysbaert B, Udry C. Development economics. A multifaceted program causes lasting progress for the very poor: evidence from six countries. Science. 2015 May 15;348(6236):1260799. doi: 10.1126/science.1260799. PMID 25977558
- [Background] Haushofer J, Shapiro J. THE SHORT-TERM IMPACT OF UNCONDITIONAL CASH TRANSFERS TO THE POOR: EXPERIMENTAL EVIDENCE FROM KENYA. Q J Econ. 2016 Nov;131(4):1973-2042. doi: 10.1093/qje/qjw025. Epub 2016 Jul 19. PMID 33087990
- [Background] Bandiera O, Robin Burgess, Narayan Das, Selim Gulesci, Imran Rasul, and Munshi Sulaiman. Labor markets and poverty in village economies. Quarterly Journal of Economics. 2017;132'(2):811-870.
- [Background] Ozer EJ, Fernald LC, Weber A, Flynn EP, VanderWeele TJ. Does alleviating poverty affect mothers' depressive symptoms? A quasi-experimental investigation of Mexico's Oportunidades programme. Int J Epidemiol. 2011 Dec;40(6):1565-76. doi: 10.1093/ije/dyr103. Epub 2011 Jul 7. PMID 21737404
- [Background] Ssewamala FM, Neilands TB, Waldfogel J, Ismayilova L. The impact of a comprehensive microfinance intervention on depression levels of AIDS-orphaned children in Uganda. J Adolesc Health. 2012 Apr;50(4):346-52. doi: 10.1016/j.jadohealth.2011.08.008. Epub 2011 Oct 26. PMID 22443837
- [Background] Plagerson S, Patel V, Harpham T, Kielmann K, Mathee A. Does money matter for mental health? Evidence from the Child Support Grants in Johannesburg, South Africa. Glob Public Health. 2011;6(7):760-76. doi: 10.1080/17441692.2010.516267. Epub 2011 May 24. PMID 20938853
- [Background] Green EP, Blattman C, Jamison J, Annan J. Does poverty alleviation decrease depression symptoms in post-conflict settings? A cluster-randomized trial of microenterprise assistance in Northern Uganda. Glob Ment Health (Camb). 2016 Feb 29;3:e7. doi: 10.1017/gmh.2015.28. eCollection 2016. PMID 28596876
- [Background] Goldman LS, Nielsen NH, Champion HC. Awareness, diagnosis, and treatment of depression. J Gen Intern Med. 1999 Sep;14(9):569-80. doi: 10.1046/j.1525-1497.1999.03478.x. PMID 10491249
- [Background] Rost K, Smith JL, Dickinson M. The effect of improving primary care depression management on employee absenteeism and productivity. A randomized trial. Med Care. 2004 Dec;42(12):1202-10. doi: 10.1097/00005650-200412000-00007. PMID 15550800
- [Background] Insel TR. Concept Clearance: NIMH's New Focus in Clinical Trials. In: NIMH; 2013.
- [Background] Angeles G, de Hoop J, Handa S, Kilburn K, Milazzo A, Peterman A; Malawi Social Cash Transfer Evaluation Team. Government of Malawi's unconditional cash transfer improves youth mental health. Soc Sci Med. 2019 Mar;225:108-119. doi: 10.1016/j.socscimed.2019.01.037. Epub 2019 Feb 15. PMID 30826585
- [Background] Weiser SD, Bukusi EA, Steinfeld RL, Frongillo EA, Weke E, Dworkin SL, Pusateri K, Shiboski S, Scow K, Butler LM, Cohen CR. Shamba Maisha: randomized controlled trial of an agricultural and finance intervention to improve HIV health outcomes. AIDS. 2015 Sep 10;29(14):1889-94. doi: 10.1097/QAD.0000000000000781. PMID 26214684
- [Background] Kim J, Ferrari G, Abramsky T, Watts C, Hargreaves J, Morison L, Phetla G, Porter J, Pronyk P. Assessing the incremental effects of combining economic and health interventions: the IMAGE study in South Africa. Bull World Health Organ. 2009 Nov;87(11):824-32. doi: 10.2471/blt.08.056580. PMID 20072767
- [Background] Nadkarni S, Genberg B, Galarraga O. Microfinance Interventions and HIV Treatment Outcomes: A Synthesizing Conceptual Framework and Systematic Review. AIDS Behav. 2019 Sep;23(9):2238-2252. doi: 10.1007/s10461-019-02443-6. PMID 30805757
- [Background] Larance L. Building social capital from the center: a village-level investigation of Bangladesh's Grameen Bank. 1998.
- [Background] Boshara R. Seven surprising findings from the asset-building field. Federal Reserve Bank of St. Louis. Bridges, Issue: Winter 2010. 2011.
- [Background] Bynner J, Paxton W. The Asset-effect. Institute for Public Policy Research; 2001.
- [Background] Fernald LC, Hamad R, Karlan D, Ozer EJ, Zinman J. Small individual loans and mental health: a randomized controlled trial among South African adults. BMC Public Health. 2008 Dec 16;8:409. doi: 10.1186/1471-2458-8-409. PMID 19087316
- [Background] Mohindra K, Haddad S, Narayana D. Can microcredit help improve the health of poor women? Some findings from a cross-sectional study in Kerala, India. Int J Equity Health. 2008 Jan 10;7:2. doi: 10.1186/1475-9276-7-2. PMID 18186918
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Glasgow RE, McKay HG, Piette JD, Reynolds KD. The RE-AIM framework for evaluating interventions: what can it tell us about approaches to chronic illness management? Patient Educ Couns. 2001 Aug;44(2):119-27. doi: 10.1016/s0738-3991(00)00186-5. PMID 11479052
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Kilburn K, Handa S, Angeles G, Tsoka M, Mvula P. Paying for Happiness: Experimental Results from a Large Cash Transfer Program in Malawi. J Policy Anal Manage. 2018 Spring;37(2):331-356. doi: 10.1002/pam.22044. Epub 2018 Feb 9. PMID 31747450
- [Background] Leichsenring F, Steinert C, Ioannidis JPA. Toward a paradigm shift in treatment and research of mental disorders. Psychol Med. 2019 Oct;49(13):2111-2117. doi: 10.1017/S0033291719002265. Epub 2019 Sep 2. No abstract available. PMID 31474241
- [Background] Cox JR, Martinez RG, Southam-Gerow MA. Treatment integrity in psychotherapy research and implications for the delivery of quality mental health services. J Consult Clin Psychol. 2019 Mar;87(3):221-233. doi: 10.1037/ccp0000370. Epub 2018 Dec 27. PMID 30589351
- [Background] Adam T, Hsu J, de Savigny D, Lavis JN, Rottingen JA, Bennett S. Evaluating health systems strengthening interventions in low-income and middle-income countries: are we asking the right questions? Health Policy Plan. 2012 Oct;27 Suppl 4:iv9-19. doi: 10.1093/heapol/czs086. PMID 23014156
- [Background] Munodawafa M, Mall S, Lund C, Schneider M. Process evaluations of task sharing interventions for perinatal depression in low and middle income countries (LMIC): a systematic review and qualitative meta-synthesis. BMC Health Serv Res. 2018 Mar 23;18(1):205. doi: 10.1186/s12913-018-3030-0. PMID 29566680
- [Background] Mill J, Davison C, Richter S, et al. Qualitative research in an international research program: Maintaining momentum while building capacity in nurses. International Journal of Qualitative Methods. 2014;13:151-169.
- [Background] Karasz A, Tofail F. Depression treatment, asset building, and household empowerment: An intervention in rural Bangladesh. In:2015.
- [Background] Bermudez LG, Ssewamala FM, Neilands TB, Lu L, Jennings L, Nakigozi G, Mellins CA, McKay M, Mukasa M. Does Economic Strengthening Improve Viral Suppression Among Adolescents Living with HIV? Results From a Cluster Randomized Trial in Uganda. AIDS Behav. 2018 Nov;22(11):3763-3772. doi: 10.1007/s10461-018-2173-7. PMID 29846836
- [Background] Banerjee S, Shamash K, Macdonald AJ, Mann AH. Randomised controlled trial of effect of intervention by psychogeriatric team on depression in frail elderly people at home. BMJ. 1996 Oct 26;313(7064):1058-61. doi: 10.1136/bmj.313.7064.1058. PMID 8898601
- [Background] Dworkin SL, Blankenship K. Microfinance and HIV/AIDS prevention: assessing its promise and limitations. AIDS Behav. 2009 Jun;13(3):462-9. doi: 10.1007/s10461-009-9532-3. Epub 2009 Mar 18. PMID 19294500
- [Background] Gonzalez JS, Batchelder AW, Psaros C, Safren SA. Depression and HIV/AIDS treatment nonadherence: a review and meta-analysis. J Acquir Immune Defic Syndr. 2011 Oct 1;58(2):181-7. doi: 10.1097/QAI.0b013e31822d490a. PMID 21857529
- [Background] Sin NL, DiMatteo MR. Depression treatment enhances adherence to antiretroviral therapy: a meta-analysis. Ann Behav Med. 2014 Jun;47(3):259-69. doi: 10.1007/s12160-013-9559-6. PMID 24234601
- [Background] Westen D, Morrison K. A multidimensional meta-analysis of treatments for depression, panic, and generalized anxiety disorder: an empirical examination of the status of empirically supported therapies. J Consult Clin Psychol. 2001 Dec;69(6):875-99. PMID 11777114
- [Background] Garcia IA, Blank AE, Eastwood EA, Karasz A. Barriers and facilitators to the implementation of SPNS interventions designed to engage and retain HIV positive women of color in medical care. AIDS Behav. 2015 Apr;19(4):655-65. doi: 10.1007/s10461-014-0837-5. PMID 25107362
- [Background] Karasz A, Bonuck K. Reducing pediatric caries and obesity risk in South Asian immigrants: randomized controlled trial of common health/risk factor approach. BMC Public Health. 2018 May 31;18(1):680. doi: 10.1186/s12889-018-5317-9. PMID 29855352
- [Background] Karasz A, Dempsey K, Fallek R. Cultural differences in the experience of everyday symptoms: a comparative study of South Asian and European American women. Cult Med Psychiatry. 2007 Dec;31(4):473-97. doi: 10.1007/s11013-007-9066-y. PMID 17985219
- [Background] Karasz A, DeSilva N, Khurshid A, K B, Ramachandran U. Contextual influences on child feeding in two South Asian immigrant groups. International Journal of Child Health and Nutrition. 2020.
- [Background] Karasz A, Jaiman A, Patel V, et al. APPLE: Development of a Lifestyle Program for South Asian Immigrant Women. Health Behavior and Policy Review. 2016;3:33-42.
- [Background] Karasz A, Margulis K, Badner V, K B. Reducing oral health risks in South Asian immigrant children: A pilot study. New York State Dental Journal. 2018;84(1):28-33.
- [Background] Karasz A, Singelis TM. Qualitative and Mixed Methods Research in Cross-cultural Psychology: Introduction to the Special Issue. J Cross Cult Psychol. 2009 Nov 1;40(6):909-916. doi: 10.1177/0022022109349172. No abstract available. PMID 21666752
- [Background] Karasz AK. Role strain and symptoms in a group of Pakistani immigrant women, City University of New York; 1998.
- [Background] Patel VV, Rajpathak S, Karasz A. Bangladeshi immigrants in New York City: a community based health needs assessment of a hard to reach population. J Immigr Minor Health. 2012 Oct;14(5):767-73. doi: 10.1007/s10903-011-9555-5. PMID 22116745
- [Background] Hamadani JD, Tofail F, Hilaly A, Mehrin F, Shiraji S, Banu S, Huda SN. Association of postpartum maternal morbidities with children's mental, psychomotor and language development in rural Bangladesh. J Health Popul Nutr. 2012 Jun;30(2):193-204. doi: 10.3329/jhpn.v30i2.11313. PMID 22838161
- [Background] Hossain SJ, Roy BR, Hossain AT, Mehrin F, Tipu SMMU, Tofail F, Arifeen SE, Tran T, Fisher J, Hamadani J. Prevalence of Maternal Postpartum Depression, Health-Seeking Behavior and Out of Pocket Payment for Physical Illness and Cost Coping Mechanism of the Poor Families in Bangladesh: A Rural Community-Based Study. Int J Environ Res Public Health. 2020 Jul 1;17(13):4727. doi: 10.3390/ijerph17134727. PMID 32630173
- [Background] Naheed A, Islam MS, Hossain SW, Ahmed HU, Uddin MMJ, Tofail F, Hamadani JD, Hussain AHME, Munir K. Burden of major depressive disorder and quality of life among mothers of children with autism spectrum disorder in urban bangladesh. Autism Res. 2020 Feb;13(2):284-297. doi: 10.1002/aur.2227. Epub 2019 Oct 24. PMID 31647184
- [Background] Pendergast LL, Scharf RJ, Rasmussen ZA, Seidman JC, Schaefer BA, Svensen E, Tofail F, Koshy B, Kosek M, Rasheed MA, Roshan R, Maphula A, Shrestha R, Murray-Kolb LE; MAL-ED Network Investigators. Postpartum depressive symptoms across time and place: structural invariance of the Self-Reporting Questionnaire among women from the international, multi-site MAL-ED study. J Affect Disord. 2014;167:178-86. doi: 10.1016/j.jad.2014.05.039. Epub 2014 Jun 12. PMID 24981251
- [Background] Desai RM, and Shareen Joshi. Can Producer Associations Improve Rural Livelihoods? Evidence from Farmer Centres in India. Journal of Development Studies. 2014;1:64-80.
- [Background] Dessai R, Joshi, S. Collective action and community development: Evidence from self-help groups in rural India. World Bank Economic Review. 2013;3(1):492-424.
- [Background] Joshi S, and Vijayendra Rao. Who Should Be at the Top of Bottom-Up Development? A Case-Study of the National Rural Livelihoods Mission in Rajasthan, India. Journal of Development Studies. 2018;54(10):1858-1877.
- [Background] Dempsey K, Karasz A. Cultural differences in health seeking for everyday symptoms. 2005.
- [Background] Karasz A, McKinley PS. Cultural differences in conceptual models of everyday fatigue: a vignette study. J Health Psychol. 2007 Jul;12(4):613-26. doi: 10.1177/1359105307078168. PMID 17584812
- [Background] Joshi S, Schultz TP. Family planning and women's and children's health: long-term consequences of an outreach program in Matlab, Bangladesh. Demography. 2013 Feb;50(1):149-80. doi: 10.1007/s13524-012-0172-2. PMID 23212440
- [Background] Joshi S, Nishtha Kochhar, and Vijayendra Rao. Are caste categories misleading? The relationship between gender and jati in three Indian states. In: Siwan Anderson LB, and Jean-Philippe Platteau, ed. Towards Gender Equity in Development. Oxford: Oxford University Press; 2018.
- [Background] Litwin AH, Jost J, Wagner K, Heo M, Karasz A, Feinberg J, Kim AY, Lum PJ, Mehta SH, Taylor LE, Tsui JI, Pericot-Valverde I, Page K; HERO Study Group. Rationale and design of a randomized pragmatic trial of patient-centered models of hepatitis C treatment for people who inject drugs: The HERO study. Contemp Clin Trials. 2019 Dec;87:105859. doi: 10.1016/j.cct.2019.105859. Epub 2019 Oct 24. PMID 31669450
- [Background] Cha ES, Kim KH, Erlen JA. Translation of scales in cross-cultural research: issues and techniques. J Adv Nurs. 2007 May;58(4):386-95. doi: 10.1111/j.1365-2648.2007.04242.x. Epub 2007 Apr 17. PMID 17442038
- [Background] Seshan G, Yang, D. Motivating migrants: A field experiment on financial decision making in transnational households. Journal of Development Economics. 2014;108:119-127.
- [Background] Carpena F, Cole, S., Shapiro, J., and Zia, B. The ABCs of financial education: experimental evidence on attitudes, behavior and cognitive biases. Management Science. 2019;65(1):346-369.
- [Background] Werner D, Bower W. Helping health workers learn: A book of methods, aids and ideas for workers at the village level. Berkeley, CA: Hesperian; 1982.
- [Background] Deaton A. The analysis of household surveys: a microeconometric approach to development policy. The World Bank Economic Review. 1997.
- [Background] Ustun TB, Chatterji S, Kostanjsek N, Rehm J, Kennedy C, Epping-Jordan J, Saxena S, von Korff M, Pull C; WHO/NIH Joint Project. Developing the World Health Organization Disability Assessment Schedule 2.0. Bull World Health Organ. 2010 Nov 1;88(11):815-23. doi: 10.2471/BLT.09.067231. Epub 2010 May 20. PMID 21076562
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Rosenberg M. Society and the adolescent self-image, revised edn. Middletown, CT: Wesleyan University. 1989.
- [Background] Beck AT, Weissman A, Lester D, Trexler L. The measurement of pessimism: the hopelessness scale. J Consult Clin Psychol. 1974 Dec;42(6):861-5. doi: 10.1037/h0037562. No abstract available. PMID 4436473
- [Background] Patrikar S, Verma A, Bhatti V, Shatabdi S. Measuring domestic violence in human immunodeficiency virus-positive women. Med J Armed Forces India. 2012 Apr;68(2):136-41. doi: 10.1016/S0377-1237(12)60020-3. Epub 2012 Apr 21. PMID 24669053
- [Background] Sherbourne CD, Stewart AL. The MOS social support survey. Soc Sci Med. 1991;32(6):705-14. doi: 10.1016/0277-9536(91)90150-b. PMID 2035047
- [Background] Lubben J, Blozik E, Gillmann G, Iliffe S, von Renteln Kruse W, Beck JC, Stuck AE. Performance of an abbreviated version of the Lubben Social Network Scale among three European community-dwelling older adult populations. Gerontologist. 2006 Aug;46(4):503-13. doi: 10.1093/geront/46.4.503. PMID 16921004
- [Background] Mason K, Smith H. Women's empowerment and social context: Resutls from five Asian Countries. In. Washington DC: World Bank; 2003.
- [Background] Govindasamy D, Ford N, Kranzer K. Risk factors, barriers and facilitators for linkage to antiretroviral therapy care: a systematic review. AIDS. 2012 Oct 23;26(16):2059-67. doi: 10.1097/QAD.0b013e3283578b9b. PMID 22781227
- [Background] Ahmed F, Arias-Granada, Y., Latif, A., Roy, D., Yanez-Pagans, M. Description of the Official Methodology used for Poverty Estimation in Bangladesh for 2016/17. Bangladesh Bureau of Statistics and World Bank Group;2017.
- [Background] Hitsman B, Buka SL, Veluz-Wilkins AK, Mohr DC, Niaura R, Gilman SE. Accuracy of a brief screening scale for lifetime major depression in cigarette smokers. Psychol Addict Behav. 2011 Sep;25(3):559-64. doi: 10.1037/a0022772. PMID 21443295
- [Background] Rubin DB, Schenker N. Multiple imputation in health-care databases: an overview and some applications. Stat Med. 1991 Apr;10(4):585-98. doi: 10.1002/sim.4780100410. PMID 2057657
- [Background] Bolker BM, Brooks ME, Clark CJ, Geange SW, Poulsen JR, Stevens MH, White JS. Generalized linear mixed models: a practical guide for ecology and evolution. Trends Ecol Evol. 2009 Mar;24(3):127-35. doi: 10.1016/j.tree.2008.10.008. PMID 19185386
- [Background] Turner EL, Prague M, Gallis JA, Li F, Murray DM. Review of Recent Methodological Developments in Group-Randomized Trials: Part 2-Analysis. Am J Public Health. 2017 Jul;107(7):1078-1086. doi: 10.2105/AJPH.2017.303707. Epub 2017 May 18. PMID 28520480
- [Background] Hemming K, Eldridge S, Forbes G, Weijer C, Taljaard M. How to design efficient cluster randomised trials. BMJ. 2017 Jul 14;358:j3064. doi: 10.1136/bmj.j3064. PMID 28710062
- [Background] Strauss AL. Qualitative analysis for social scientists. In:1987:319.
- [Background] Karasz A, Anne S, Hamadani JD, Tofail F. The ASHA (Hope) Project: Testing an Integrated Depression Treatment and Economic Strengthening Intervention in Rural Bangladesh: A Pilot Randomized Controlled Trial. Int J Environ Res Public Health. 2021 Jan 1;18(1):279. doi: 10.3390/ijerph18010279. PMID 33401489
- [Background] Campbell M.J. W, S. J. . How to Design, Analyses and Report Cluster Randomized Trials in Medicine and Health Related Research. New York: Wiley; 2014.
- [Background] Shea MT, Elkin I, Imber SD, Sotsky SM, Watkins JT, Collins JF, Pilkonis PA, Beckham E, Glass DR, Dolan RT, et al. Course of depressive symptoms over follow-up. Findings from the National Institute of Mental Health Treatment of Depression Collaborative Research Program. Arch Gen Psychiatry. 1992 Oct;49(10):782-7. doi: 10.1001/archpsyc.1992.01820100026006. PMID 1417430
- [Background] Donner A, Klar, N. Design and Analysis of Cluster Randomization Trials in Health Research. London: Arnold; 2000.
- [Background] Rahman A, Malik A, Sikander S, Roberts C, Creed F. Cognitive behaviour therapy-based intervention by community health workers for mothers with depression and their infants in rural Pakistan: a cluster-randomised controlled trial. Lancet. 2008 Sep 13;372(9642):902-9. doi: 10.1016/S0140-6736(08)61400-2. PMID 18790313
- [Background] Swartz HA, Grote NK, Graham P. Brief Interpersonal Psychotherapy (IPT-B): Overview and Review of Evidence. Am J Psychother. 2014;68(4):443-62. doi: 10.1176/appi.psychotherapy.2014.68.4.443. PMID 26453346
- [Background] Onken LS, Carroll KM, Shoham V, Cuthbert BN, Riddle M. Reenvisioning Clinical Science: Unifying the Discipline to Improve the Public Health. Clin Psychol Sci. 2014 Jan 1;2(1):22-34. doi: 10.1177/2167702613497932. PMID 25821658
- [Background] Riddle M, Clark D. Behavioral and social intervention research at the National Institute of Dental and Craniofacial Research (NIDCR). J Public Health Dent. 2011 Winter;71 Suppl 1:S123-9. doi: 10.1111/j.1752-7325.2011.00216.x. No abstract available. PMID 21656969